CLINICAL TRIAL: NCT00009568
Title: Platelet Dysfunction in Patients Treated With SSRI Versus Non-SSRI Antidepressants
Brief Title: Platelet Function in Patients Treated With SSRI and Non-SSRI Antidepressants
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 010077; 01-CC-0077
Record Dates: First submitted 2001-02-01; First posted 2001-02-02 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-01

CONDITIONS: Depression
Keywords: Antidepressants; Platelet Function; SSRI; Depression; Bleeding Time
MeSH Terms: conditions — Depression

SUMMARY:
This study will examine the effect of a class of antidepressant medications called selective serotonin reuptake inhibitors (SSRIs) on platelet function. Platelets are small blood cells that help stop bleeding after injury to a blood vessel by forming a clot, or plug, in the vessel. Some medications impair platelet function, leading to increased bruising and bleeding. SSRIs decrease an important platelet component called serotonin, which may cause bleeding in some patients. SSRIs include fluoxetine (Prozac), sertraline (Zoloft), paroxetine (Paxil), fluvoxamine (Luvox) and citalopram (Celexa).

Patients 18 years of age and older being treated for depression with a SSRI or the non-SSRI bupropion (Wellbutrin) may be eligible for this study. Subjects will be recruited from a private clinic in Washington, D.C.

Participants will provide a history of their current medications and past history of bleeding. They will have about 4 tablespoons of blood drawn for tests to measure blood cell counts and platelet function. The study takes about 1 hour. The results of the SSRI-treated group and the bupropion-treated group will be analyzed and compared.

This study may provide information that will help health care providers make treatment decisions to minimize possible adverse effects of medications in patients with depression.

DETAILED DESCRIPTION:
This study will evaluate platelet function in patients during treatment with selective serotonin reuptake inhibitors (SSRIs) which are widely used antidepressant agents. SSRIs, which are known to decrease platelet serotonin content, have been reported to be associated with bleeding in a minority of patients and recently have been associated with an increase in gastrointestinal bleeding. The purpose of this study is to better understand the potential risks of bleeding associated with mild platelet dysfunction in patients using SSRIs and to determine whether a global test of platelet function, as performed on the platelet function analyzer-100, is able to identify the changes in platelet function associated with SSRI use. Until recently, platelet function testing has utilized platelet aggregation studies which are very labor-intensive and require highly skilled technicians; a newer instrument, the Platelet Function Analyzer-100 (PFA-100, Dade Behring, Deerfield, IL) requires much less technical input to evaluate platelet function. The patients will be selected from a private clinic in the Washington, DC, area and will undergo a baseline assessment (history of bleeding and/or thrombosis), blood tests for routine blood counts, chemistries, and platelet function using the PFA-100. The analysis will include a statistical comparison of the platelet function in patients on SSRIs with those on a non-SSRI antidepressant medication (bupropion). It will also include an analysis of the results of the PFA-100 compared to the results of platelet aggregation. The results of the study may provide a better understanding of platelet function and screening for platelet function defects in patients using SSRIs.

ELIGIBILITY:
INCLUSION CRITERIA:

Male or female subjects with a diagnosis of depression over the age of 18 years,

Subjects currently prescribed and taking a stable dose of SSRI for at least 6 weeks, or

Subjects currently prescribed and taking a stable dose of bupropion for at least 6 weeks.

EXCLUSION CRITERIA:

Inherited or acquired coagulopathies or platelet disorders

Abnormal thyroid function (TSH less than 0.42 or greater than 4.4 micro IU/ml and free T4 less than 1.0 or greater than 1.9 ng/dL).

Severe depression as indicated by the following: Major depressive disorder single episode, severe without psychotic features DSM-IV 296.23; Major depressive disorder single episode, severe with psychotic features DSM-IV 296.24; Major depressive disorder recurrent, severe without psychotic features DSM-IV 296.33; Major depressive disorder recurrent, severe with psychotic features DSM-IV 296.34.

Patients who are currently receiving coumadin or heparin, non-steroidal antiinflammatory drugs (NSAIDs), acetylsalicylic acid (Aspirin), corticosteroids, chemotherapy, or other medications known to interfere with platelet function studies will not be eligible.

Patients taking NSAIDS and aspirin or other medications known to interfere with platelet function studies will be eligible if they discontinue these medications for more than 10 days prior to testing.

Patients who are taking the following psychotropic medications: valproic acid, carbamazepine, buspiron, atypical antipsychotics, or any other psychotropic medications will not be eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70
Dates: Start 2001-01; Study Completion 2005-01

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Alderman CP, Moritz CK, Ben-Tovim DI. Abnormal platelet aggregation associated with fluoxetine therapy. Ann Pharmacother. 1992 Dec;26(12):1517-9. doi: 10.1177/106002809202601205. PMID 1482806
- [Background] Berk M, Jacobson BF, Hurly E. Fluoxetine and hemostatic function: a pilot study. J Clin Psychiatry. 1995 Jan;56(1):14-6. PMID 7836333